CLINICAL TRIAL: NCT01533558
Title: Pharmacokinetics of Caspofungin (Cancidas ®) Given Intravenously as Therapy to Patients With an Invasive Fungal Infection in the Intensive Care Unit - a Search for Co-variates
Acronym: CASCADE
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: AKF UMCN 11.02
Record Dates: First submitted 2012-01-19; First posted 2012-02-15 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Invasive Fungal Infection
Keywords: caspofungin; pharmacokinetics; invasive fungal infection; candidiasis; aspergillosis; intensive care
MeSH Terms: conditions — Invasive Fungal Infections; Candidiasis; Aspergillosis | interventions — Caspofungin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples for determination of caspofungin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- caspofungin: caspofungin dosing
  Interventions: Drug: caspofungin

INTERVENTIONS:
Drug: caspofungin — normal dosage for caspofungin, not adapted for the study
  Other Names: Cancidas

SUMMARY:
The pharmacokinetics of caspofungin are expected to be different in ICU patients compared to non-ICU patients. The investigators will determine caspofungin concentrations in 20 ICU patients, who will get caspofungin as standard care.

Full PK curves will be taken on day 3 and a limited PK curve on day 7, trough levels will be taken daily.

DETAILED DESCRIPTION:
The pharmacokinetics of caspofungin are expected to be different in ICU patients compared to non-ICU patients and healthy volunteers due to underlying disease(s). Therefore, extrapolation of data from healthy volunteers and non-ICU patients is not possible.

To be able to include 20 patients within the study duration, a multi-centre approach is necessary.

Patients will receive standard care, as stated in the SPC or according to local protocols. Blood sampling for PK analysis will be retrieved through a central venous catheter. Approximately 60mL will be drawn in total for this study. Patients will be monitored daily during the treatment period for adverse events of the study drug.

Although steady state of caspofungin will be achieved after approximately 14 days of treatment, full PK curves will be taken on day 3. As probably not all patients included will be treated with caspofungin for 14 days, taking full PK curves on day 14 is considered not feasible. These two moments of PK analysis will enable the determination steady state and enable the determination of intra-individual variability.

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted to an ICU
* Subject is at least 18 and not older than 65 years of age on the day of the first dosing
* Subject has been treated with caspofungin for a maximum of two days before enrolment in this trial
* Is managed with a central venous catheter

Exclusion Criteria:

* Is known to be hypersensitive to echinocandin antifungal agents
* Documented history of sensitivity to medicinal products or excipients similar to those found in the caspofungin preparation
* Positive HIV test or hepatitis B or C test
* History of QT time prolongation
* History of or current abuse of drugs, alcohol or solvents
* Has previously participated in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care patients with invasive fungal infection
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | day 3 and day 7
  AUC0-tau, AUC0-inf (Time Frame: predose, 0.5, 1, 2, 4, 6, 8, 12, 16, 20 and 24 hours post-dose on Day 3 and predose, 1, 4, 8, 12 hours + 6 days after the dose on Day 7) of caspofungin

SECONDARY OUTCOMES:
co-variates influencing PK of caspofungin | day 3 and day 7
  identify co-variates of influence on the pharmacokinetics of caspofungin
Number of Participants with Adverse Events | 14 days
  the adverse events will be recorded in IC patients during the study

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brüggemann, PhD, PharmD, Principal Investigator — Radboud University Medical Center
Locations (4):
- Netherlands (4):
  - Rijnstate Hospital, Arnhem
  - Canisius Wilhelmina Hospital (CWZ), Nijmegen
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - University Medical Centre Utrecht, Utrecht

REFERENCES:
- [Result] Muilwijk EW, Schouten JA, van Leeuwen HJ, van Zanten AR, de Lange DW, Colbers A, Verweij PE, Burger DM, Pickkers P, Bruggemann RJ. Pharmacokinetics of caspofungin in ICU patients. J Antimicrob Chemother. 2014 Dec;69(12):3294-9. doi: 10.1093/jac/dku313. Epub 2014 Aug 19. PMID 25139840